CLINICAL TRIAL: NCT05123235
Title: The Effectiveness of a Telehealth-Based Physical Activity Intervention in Adolescents Receiving Treatment for Obesity
Brief Title: Effectiveness of a Telehealth-based Physical Activity Intervention
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: After starting to recruit it became apparent that the participants did not want to participate in a telehealth intervention.
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-001684
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Physical Inactivity; Obesity, Childhood
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Physical activity group and a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): The intervention will last 11 weeks, and participants in the intervention group will have individual weekly web-meeting using a video conferencing platform. The weekly meeting is expected to last approximately 30 minutes. During this meeting, participants will report on the past week's physical activity goals, failures and successes, set goals for the next week, discuss that week's behavioral strategy to promote physical activity for that week, and engage around 5 minutes of physical activity. The topics that will be discussed in the newsletters and weekly meetings will include behavioral strategies for physical activity changes. Those in the control group will also be contacted weekly for 11 weeks and will be asked about their physical activity levels for the past week. These meetings will also occur using video conferencing and last 5 minutes.
  Interventions: Behavioral: Physical Activity
- Control (No Intervention): During the 11 weeks the participants in the control group will have a weekly check in meeting using a video conferencing platform. The weekly meeting is expected to last approximately 5 minutes. During this meeting, participants will report on the past week's physical activity levels.

INTERVENTIONS:
Behavioral: Physical Activity — the participants will be encouraged to set their own physical activity goals weekly and using behavioral strategies work towards meeting those goals. The behavioral strategies will be discussed weekly for 30 minutes a telehealth method.
  Arms: Physical Activity

SUMMARY:
This study is a 11 week telehealth intervention focusing on increasing physical activity in adolescents who are receiving medical care for obesity. The participants will be randomized into two groups: control and intervention. During the 11 weeks both groups will be contacted once a week for a video call. The control group will report their past week physical activity levels and the intervention group will review the material in weekly newsletters on behavior changes related to physical activity. Physical activity levels will be measures before and after the intervention.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a physical activity telehealth intervention will increase the amount of moderate-to-vigorous physical activity among 14-17 year olds who are receiving obesity treatment. A secondary purpose is to determine if a telehealth physical activity intervention will impact the adolescents' body mass index (BMI) z-score who are receiving treatment for obesity. The participants will complete questionnaires to measure current physical activity levels, physical activity enjoyment, motivation, and strategies to be active. The study investigators will also review the participants medical records to get BMI. Participants will be randomized into either an intervention or standard care control group at a 1:1 ratio (intervention-control). A computer-generated randomization list will be created by an individual not associated with the study. The intervention will last 11 weeks, and participants in the intervention group receive standard medical care and will have individual weekly web-meeting using a video conferencing platform, Microsoft Teams. The weekly meeting is expected to last approximately 30 minutes. During this meeting, participants will report on the past week's physical activity goals, failures and successes, set goals for the next week, discuss that week's behavioral strategy to promote physical activity for that week, and engage around 5 minutes of physical activity. The topics that will be discussed in the newsletters and weekly meetings will include behavioral strategies for physical activity changes. Those in the control group will also receive standard medical care and be contacted weekly for 11 weeks and will be asked about their physical activity levels for the past week. These meetings will also occur using video conferencing and last 5 minutes. After a regular visit to the medical clinic (6 weeks from the 1st study visit) the study investigators will review medical records from all participants for height, weight, and BMI. About 12 weeks after the 1st study visit, during a regular clinic visit all participants will complete questionnaires to measure current physical activity levels, physical activity enjoyment, motivation, and strategies to be active. The study investigators will also review the participants medical records to get height, weight and BMI.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years of age
* receiving treatment for obesity
* have a smart device for video conferencing

Exclusion Criteria:

* under 14 years of age
* Pregnant
* Type 1 or Type 2 Diabetes
* Neuromuscular disease that impacts moving
* Parent or child unable to speak or write in English.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity participation | weeks 1 and 12
  minutes spent in physical activity
Change in BMI z-score | weeks 1, 6, and 12
  BMI z-score will be calculated from BMI and CDC normative data
Change in BMI percentile | weeks 1, 6, and 12
  BMI percentile will be calculated from BMI and CDC normative data

SECONDARY OUTCOMES:
Change in physical activity enjoyment | weeks 1 and 12
  physical activity enjoyment scale - Likert rating from 1-5 a higher total summary score means more enjoyment
Change in physical activity motivation | weeks 1 and 12
  motivation to exercise scale, Likert scale 1-5 where 1=not very true for me to 5=very true for me; 5 different subscales are calculated: amotivation, external regulation, introjected regulation, identified regulation, and intrinsic motivation
Change in physical activity strategies | weeks 1 and 12
  physical activity self management questionnaire, Likert scale 1-5 where 1=not very often to 5=very often. A higher score means that the person uses more posititve self management strategies to engage in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Katrina D DuBose, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No